CLINICAL TRIAL: NCT02464137
Title: A Phase I Trial of Stereotactic HYpofractionateD RadioAblative (HYDRA) Treatment of Advanced Laryngeal Cancer
Brief Title: HYpofractionateD RadioAblative (HYDRA) Treatment of Advanced Laryngeal Cancer
Acronym: HYDRA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: unexpected toxicities
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 052014-085
Record Dates: First submitted 2015-05-07; First posted 2015-06-08 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-03

CONDITIONS: Squamous Cell Carcinoma of the Larynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation (Experimental): Patients in each dose cohort will all be treated as a single group. The starting dose will be 8.5 Gy per fraction for 5 fractions (total dose = 42.5 Gy). Subsequent cohorts of patients will receive an additional 0.5 Gy per fraction.
  Interventions: Radiation: radiation

INTERVENTIONS:
Radiation: radiation — Patients in each dose cohort will all be treated as a single group. The starting dose will be 8.5 Gy per fraction for 5 fractions (total dose = 42.5 Gy). Subsequent cohorts of patients will receive an additional 0.5 Gy per fraction.
  Other Names: HYpofractionateD RadioAblative

SUMMARY:
single-modality phase I dose escalation toxicity study for first-line curative treatment of head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
HYDRA will consist of 5 fraction SBRT treatment targeting only grossly evident disease localized by examination and standard diagnostic CT, MR, and PET-CT imaging. Prophylactic coverage of uninvolved at-risk mucosal and nodal drainage basins will be strictly disallowed. The initial dose cohort will be treated to a total of 42.5 Gy in five equal fractions delivered every other day over a two week period (biologically equivalent to 66 Gy delivered in 2 Gy daily fractions), drawn from our successful institutional experience with similar dosing and fractionation for early-stage larynx SBRT. Escalation of total dose will proceed in 2.5 Gy increments, up to a final target dose of 50 Gy.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age with histologically proven squamous cell carcinoma of the larynx.
* Stage T1-2N1-2c/T3-4N0-2c disease, as defined by American Joint Committee on Cancer (AJCC) criteria.
* ECOG (Zubrod) performance status 0-2.
* Must be functionally and technically fit for partial laryngectomy.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy.
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients who have undergone resection of primary disease.
* Patients who have received induction chemotherapy for their cancer diagnosis.
* Patients who have undergone a diverting tracheostomy which is either a) traversing directly through tumor, b) has been placed for true airway insufficiency. Patients with a tracheostomy placed preemptively for impending airway compromise remain eligible for enrollment.
* Prior cancer diagnosis, except appropriately treated localized epithelial skin cancer or cervical cancer.
* Prior radiation therapy to the head and neck region.
* Women of childbearing potential (a woman of child-bearing potential is a reproductively mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months [i.e., who has had menses at any time in the preceding 24 consecutive months]) and male participants must practice effective contraception (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study.
* Patients unable or unwilling to give written, informed consent.
* Severe, active co-morbidity, defined as follows:

  1. Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months.
  2. Transmural myocardial infarction within the last 6 months.
  3. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration.
  4. Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before registration.
  5. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol.
  6. Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. Protocol-specific requirements may also exclude immuno-compromised patients.
  7. History of treatment with potent immunosuppressive drugs for such conditions as post organ transplant, severe rheumatoid arthritis, etc. within the past 6 months.
* Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants
* Evidence of metastatic disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-04-27 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
toxicities | 90 days
  Number of participants with acute related serious adverse events

SECONDARY OUTCOMES:
adverse events | 2 years
  Number of participants with adverse events
quality of life | 5 years
  Scale of quality of life questionnaire
disease control | 5 years
  Number of participants with disease control (no evidence of disease, progression)
dosimetric improvement | 2 weeks
  Scores of radiation quality review

CONTACTS AND LOCATIONS:
Overall Officials: Lucien Nedzi, MD, Principal Investigator — UTSW Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States